CLINICAL TRIAL: NCT01076920
Title: Administration of Mesenchymal Stem Cells in Patients With Chronic Ischemic Cardiomyopathy
Brief Title: Mesenchymal Stem Cells and Myocardial Ischemia
Acronym: MESAMI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: French Blood Establishment (Other); Nantes University Hospital (Other); Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0505008
Record Dates: First submitted 2010-02-10; First posted 2010-02-26 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Chronic Myocardial Ischemia; Left Ventricular Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Left

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention arm (Experimental)
  Interventions: Genetic: Mesenchymal stem cells

INTERVENTIONS:
Genetic: Mesenchymal stem cells — 60x106 MSCs Trans-endocardial intramyocardial injections (n=14-16)

SUMMARY:
Ischemic cardiomyopathies are a leading cause of death in both men and women. When a person has a heart attack, blood is unable to reach a certain area of the heart, and if the blood supply is not re-established quickly, that area of the heart can suffer permanent damage. While recovery from a heart attack can be managed through medications and lifestyle changes, these treatments can not reverse the all damage to the heart. Current research is focusing on the development of cell-based therapies using stem cells to repair organs that have been irreversibly damaged by disease. A specific form of stem cells, called adult mesenchymal stem cells (MSCs), has shown promise for heart repair. This study will evaluate the safety of injecting MSCs directly into the heart to repair and restore heart function in people who have had a heart attack and who have chronic myocardial ischemia with heart failure.

DETAILED DESCRIPTION:
Mesenchymal stem cells from the bone marrow can differentiate into endothelial cells and participate in the development of new blood vessels in ischemic tissue. The aim of the study is in a phase I safety study to evaluate the clinical effect of autologous mesenchymal stem cell therapy in patients with severe chronic myocardial ischemia.10 patients with reversible ischemia on a SPECT will be treated with direct intramyocardial injections of autologous isolated and expanded mesenchymal stem cells.Clinical and objective evaluations will be performed at baseline and during 24 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75
2. Male or female
3. NYHA (Heart failure) Class II-IV or Angina pectoris CCS Class III or IV or symptoms consistent with)
4. Chronic coronary artery disease with left ventricular function below 35%
5. Stable medical therapy for at least one month
6. Reversible perfusion defects by SPECT
7. Not a candidate for coronary artery by-pass surgery due to poor targets or small vessels and not a candidate for percutaneous intervention due to small vessels or unreachable coronary lesions due to complicated anatomy
8. Implantable Cardiovertor Defibrillator

Exclusion Criteria:

1. Acute coronary syndrome, revascularization (PCI or CABG), or cardiac resynchronization during the last 3 months
2. Sustained ventricular
3. Further revascularization planned for the next 30 days.
4. Chronic atrial fibrillation.
5. A wall thickness in the target region <8 mm as determined by 2D echocardiography (the target region is defined at the time of NOGA® mapping).
6. An LV thrombus.
7. Severe peripheral vascular disease precluding femoral artery access as determined at time of original catheterization.
8. Aortic stenosis as determined as valve area less than 1 cm2 that prohibits catheter access to the LV.
9. Human immunodeficiency virus (HIV1-2), HTLV-1 and 2.
10. An active uncontrolled infection.
11. A prosthetic aortic valve.
12. A current or prior history within the last 3 years of neoplasm (excluding basal cell) and/or any active neoplasm within the last 24 months.
13. Pregnancy or breastfeeding.
14. Active participation in other research therapy for cardiovascular repair/regeneration.
15. Any medical condition that would affect the investigator's ability to evaluate the subject's condition or could compromise the subject's safety.
16. Any condition that, in the judgment of the investigator, would prohibit the subject from participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-10; Primary Completion 2014-02 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Evaluate safety and feasibility of transendocardial injection using the NogaStar XP Mapping Catheter with the MyostarTM Left Ventricular Injection Catheter of autologous MSC in subjects with chronic myocardial ischemia and left ventricular dysfunction | 30 days

SECONDARY OUTCOMES:
Change from baseline in SF-36, VO2max, 6 min walk test, and the NYHA, CCS Classifications Effect related to cardiac function | 30 days to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: jerome RONCALLI, MD, PhD, Principal Investigator — University Hospital Of TOULOUSE
Locations (1):
- University Hospital (Rangueil), Toulouse, France

REFERENCES:
- [Derived] Guijarro D, Lebrin M, Lairez O, Bourin P, Piriou N, Pozzo J, Lande G, Berry M, Le Tourneau T, Cussac D, Sensebe L, Gross F, Lamirault G, Huynh A, Manrique A, Ruidavet JB, Elbaz M, Trochu JN, Parini A, Kramer S, Galinier M, Lemarchand P, Roncalli J. Intramyocardial transplantation of mesenchymal stromal cells for chronic myocardial ischemia and impaired left ventricular function: Results of the MESAMI 1 pilot trial. Int J Cardiol. 2016 Apr 15;209:258-65. doi: 10.1016/j.ijcard.2016.02.016. Epub 2016 Feb 2. PMID 26901787